CLINICAL TRIAL: NCT07021937
Title: Investigating Brain PLASTICity and GLP-1 Receptor Agonists in the Treatment of Obesity: The PLASTIC Trial
Brief Title: Brain Plasticity and GLP-1 Receptor Agonist Treatment for Obesity
Acronym: PLASTIC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Minnesota (Other); The Metis Foundation (Other)
Responsible Party: Principal Investigator, Allison Shapiro, Assistant Professor, University of Colorado, Denver
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pending; Pending (Other: Pending)
Record Dates: First submitted 2025-06-03; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Obesity/Therapy
Keywords: adolescent; adult; brain function; glucagon-like peptide-1 receptor agonists; eating behaviors; appetite sensations
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — semaglutide; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: study statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Pubertal Adolescent - Continuous Treatment (Experimental): Pubertal adolescents defined as Tanner stage 2-4 and/or 12-15 y/o who will receive 32 weeks of semaglutide (s.c.)
  Interventions: Drug: Semaglutide 1.7mg subcutaneous
- Pubertal Adolescent - Early Treatment Cessation (Experimental): Pubertal adolescents defined as Tanner stage 2-4 and/or 12-15 y/o who will receive 24 weeks of semaglutide (s.c.) followed by 8 weeks of placebo
  Interventions: Drug: Semaglutide 1.7mg subcutaneous; Drug: Placebo
- Post-Pubertal Adolescent - Continuous Treatment (Experimental): Post-pubertal adolescents defined as Tanner stage 5 and/or 16-18 y/o who will receive 32 weeks of semaglutide (s.c.)
  Interventions: Drug: Semaglutide 1.7mg subcutaneous
- Post-Pubertal Adolescent - Early Treatment Cessation (Experimental): Post-pubertal adolescents defined as Tanner stage 5 and/or 16-18 y/o who will receive 24 weeks of semaglutide (s.c.) followed by 8 weeks of placebo
  Interventions: Drug: Semaglutide 1.7mg subcutaneous; Drug: Placebo
- Adult - Continuous Treatment (Active Comparator): Adults defined as 30-45 y/o who will receive 32 weeks of semaglutide (s.c.)
  Interventions: Drug: Semaglutide 1.7mg subcutaneous
- Adult - Early Treatment Cessation (Active Comparator): Adults defined as 30-45 y/o who will receive 24 weeks of semaglutide (s.c.) followed by 8 weeks of placebo
  Interventions: Drug: Semaglutide 1.7mg subcutaneous; Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide 1.7mg subcutaneous — Semaglutide subcutaneous max dose of 1.7mg over 24 or 32 weeks of active treatment
  Other Names: SEMA
Drug: Placebo — Placebo saline solution subcutaneous
  Arms: Adult - Early Treatment Cessation; Post-Pubertal Adolescent - Early Treatment Cessation; Pubertal Adolescent - Early Treatment Cessation

SUMMARY:
Glucagon-like peptide 1 receptor agonists (GLP-1RA), such as Ozempic and Wegovy, have been rapidly adopted for the treatment of obesity in both youth and adults. However, despite this rapid adoption and the known GLP-1RA mechanism of action for weight loss, which targets brain circuits responsible for appetite and eating behaviors, almost nothing is known about how these drugs affect the brain in youth who are treated for obesity, or how these drugs affect the brain of youth differently from adults. The goal of the current study is to compare youth and adults with obesity who are treated a GLP-1RA and measure potential difference in GLP-1RA associated change in brain function, appetite, and eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* male or female (sex assigned at birth)
* 12-18 y/o with obesity (BMI>120% of the 95th %ile)
* 30-45 y/o with obesity (BMI>35 kg/m2)

Exclusion Criteria:

* treated with glucagon-like peptide-1 (GLP-1) agonists (e.g., exenatide, liraglutide, semaglutide, tirzepatide) for weight management in the prior 3 months
* currently taking anti-psychotic medications (anti-depressants accepted)
* diagnosis of type 2 diabetes
* current or lifetime anorexia nervosa or current bulimia nervosa
* head injury resulting in loss of consciousness >30min
* neurological disorder (e.g., Parkinson's disease) or history of stroke
* any contraindication to receiving a MRI (e.g., orthodontal braces)
* psychological/behavioral dysfunction (e.g., autism spectrum disorder) or physical impairment that would interfere with study procedures, as determined by study physician
* if female, desiring to become pregnant, or currently pregnant or breastfeeding

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2031-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
hypothalamic functional activation | From enrollment to the end of trial at 32 weeks
  blood oxygen-level dependent signal via resting-state functional magnetic resonance imaging
hypothalamic functional connectivity | From enrollment to the end of trial at 32 weeks
  blood oxygen-level dependent signal via resting-state functional magnetic resonance imaging
ad libitum food intake | From enrollment to the end of trial at 32 weeks
  Measured as kcal consumed from standardized ad libitum meal
appetite sensations | From enrollment to the end of trial at 32 weeks
  pre- and post-meal hunger, desire to eat, amount feel can eat, and fullness

CONTACTS AND LOCATIONS:
Overall Officials: Allison Shapiro, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Pending consent authorization by participants